CLINICAL TRIAL: NCT05857982
Title: A Prospective, Open-label, Single-arm Clinical Study of Mitoxantrone Hydrochloride Liposome Injection Combined With Daratumumab and Dexamethasone in the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK2023022-IR01
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This study is a single-arm trial with ORR as the main endpoint. Due to limited data on mitoxantrone hydrochloride liposome injection, no statistical hypothesis will be made in this study to ensure the accuracy of the estimate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDD group (Experimental): Dexamethasone 20 mg/d, on the same day of daratumumab injection; Mitoxantrone hydrochloride liposome injection: 20 mg/m2, d1; Daratumumab: 16 mg/Kg, once a week for the first 8 weeks; then changed to once every two weeks; Each cycle is 4 weeks long and the maximum number of cycles is 6.
  Interventions: Drug: Mitoxantrone hydrochloride liposome/Dexamethasone/daratumumab

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome/Dexamethasone/daratumumab — Dexamethasone 20 mg/d, on the same day of daratumumab injection; Mitoxantrone hydrochloride liposome injection: 20 mg/m2, d1; Daratumumab: 16 mg/Kg, once a week for the first 8 weeks; then changed to once every two weeks; Each cycle is 4 weeks long and the maximum number of cycles is 6.
  Other Names: Mitoxantrone hydrochloride liposome

SUMMARY:
A prospective, open-label, single-arm clinical study of mitoxantrone hydrochloride liposome injection combined with daratumumab and dexamethasone in the treatment of relapsed/refractory multiple myeloma

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-arm study. It is expected to include 20 patients with relapsed/refractory multiple myeloma who will receive combined treatment. The recommended dose of mitoxantrone hydrochloride liposome injection is 20mg/m2 (the dose can be adjusted according to the patient's tolerance, but the minimum dose is not less than 12mg/m2). Each cycle is 4 weeks long and the maximum number of cycles is 6.

Dexamethasone 20 mg/d, on the same day of daratumumab injection; Mitoxantrone hydrochloride liposome injection: 20 mg/m2, d1; Daratumumab: 16 mg/Kg, once a week for the first 8 weeks; then changed to once every two weeks; The study includes a screening period (within 28 days), a treatment period (up to 6 cycles), and a follow-up period (safety follow-up, survival follow-up, planned for 2 years).

The subjects signed an informed consent form and underwent baseline examination during the screening period. Eligible patients were enrolled in the treatment period. All subjects underwent relevant examinations as stipulated in the protocol during the treatment process to observe efficacy and safety. After the treatment period ends, they will enter the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age :18-75 years, male or female; 2. Meet the definition of relapsed/refractory multiple myeloma; 3. At least one of the following can be evaluated:

  1. Blood M protein level ≥10g/L;
  2. 24-hour urine M protein level ≥200mg;
  3. The difference between involved and uninvolved serum free light chain (dFLC) ≥100mg/L;
  4. Extramedullary lesions with a diameterday≥2cm; 4. ECOG score 0-2 points; 5. Laboratory tests meet the following criteria:

  <!-- -->

  1. Absolute neutrophil count (ANC) ≥1.0x109/L;
  2. Platelets (PLT) ≥50x109/L;
  3. Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN);
  4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN;
  5. Creatinine clearance rate (Ccr) ≥30ml/min.

Exclusion Criteria:

* 1.Expected survival time <3 months. 2.History of allergy to mitoxantrone or liposomal drugs; previous treatment with mitoxantrone or other anthracycline therapy, total cumulative dose of mitoxantrone >360 mg/m2 (other anthracycline drugs are equivalent to 1mg mitoxantrone, 2mg doxorubicin or 0.5mg epirubicin).

  3.Impaired cardiac function or significant heart disease, including but not limited to: a) Myocardial infarction or viral myocarditis within 6 months before screening. b) Existing heart disease requiring treatment at the time of screening, such as unstable angina pectoris, chronic congestive heart failure (NYHA≥2), arrhythmia, valve disease, etc., or persistent myocardial disease. c) QTc interval>480ms at screening or long QTc syndrome. d) Ejection fraction less than 50% at screening or lower than the lower limit of the study center's examination value range.

  4.HBsAg or HBcAb positive and HBV-DNA titer higher than the lower limit of the study center's detection value, or HCV antibody positive and HCV-RNA titer higher than the lower limit of the study center's detection value, or HIV antibody positive.

  5.Bacterial infection, fungal infection or viral infection requiring systemic treatment within 1 week before administration of the study drug.

  6.Pregnant or lactating women. 7.Other situations judged by investigator as inappropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective response rate (ORR): Objective response includes partial response (PR), very good partial response (VGPR), complete response (CR), and strictly defined complete response (sCR).

SECONDARY OUTCOMES:
Adverse Eventsl | 6 months
  hematological and non-hematologica Adverse Eventsl (NCI CTCAE v5.0);
DoR | 1 year
  Duration of response (DoR)
1-year PFS rate | 1 year
  1-year progression-free survival rate (PFS)
1-year PFS OS | 1 year
  1-year overall survival rate (OS)
1-year extramedullary relapse rate. | 1 year
  1-year extramedullary relapse rate.

CONTACTS AND LOCATIONS:
Overall Officials: Bingzong LI, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China